CLINICAL TRIAL: NCT03680066
Title: Assessing Tolerance to "May Contain Traces" Processed Foods in Tree Nuts or Peanut Allergic Children.
Brief Title: Study to Assess Tolerance of Traces in Peanut/Tree Nut Allergic Children.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment stopped due to low number of subjects
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Philippe Eigenmann, Head, Pediatric Allergy Unit, Department of Pediatrics, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCER 2017-01413
Record Dates: First submitted 2018-07-25; First posted 2018-09-21 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Food Allergy; Peanut Allergy; Tree Nut Allergy
Keywords: Peanut allergy; Tree Nut allergy; Precautionary allergen labeling; May contain traces; Allergen threshold
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Nut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foods with traces (Experimental): Oral food challenge with foods with traces
  Interventions: Other: Oral food challenge to foods with traces

INTERVENTIONS:
Other: Oral food challenge to foods with traces — Subjects will undergo an open food challenge to 3 processed foods labeled with "may contain traces". The following foods (similar for all patients) will be given in one dose in the size of a regular serving:
  * cookies, max 30 g;
  * chocolate, max 30 g;
  * breakfast cereals, max 50 g.
  Each meal will be administered with a 1 hour observation period in between and at the end.

SUMMARY:
This protocol will help better define whether patients with peanut and/or tree nut food allergy can tolerate traces in products with precautionary allergen labelling.

DETAILED DESCRIPTION:
Visit 1 (V1): During this visit at the Pediatric Research Platform at the Children's Hospital, subjects will undergo an open food challenge to 3 processed foods labeled with "may contain traces" by following safety and accuracy guidelines for food challenges (7). The following foods (similar for all patients) will be given in one dose in the size of a regular serving:

* cookies, max 30 g;
* chocolate, max 30 g;
* breakfast cereals, max 50 g.

Each meal will be administered with a 1 hour observation period in between and at the end.

If the patient does not react to any of the foods or has only oral itching (mild symptoms), he/she will be instructed to stop the ban on "may contain" foods and eat them regularly. If the patient has more than mild symptoms, the study will be stopped and the patient will be banned from eating foods with traces. The study subjects with a negative challenge and instructed to eat foods with the "may contain" label will be provided emergency medications and instruction on when and how to use them according to current guidelines (8).

An age appropriate quality of life questionnaire will be filled out by the parents/patient during the visit.

For the following 3 months after "may contain food" challenges, the patients will be invited to eat on a regular basis any foods labeled as "may contain" tree nuts and/or peanuts and record the consumption on a diary. Such foods will only be eaten in presence of a family member instructed for the measures to be taken in case of a reaction. They will record any history of reaction and contact the study team. The brand name of the food, and if available the batch will be recorded. The participants will store the study food and its packaging safely in a box and bring it along at V2 for allergen content analysis.

If a reaction occurs, the food will be analyzed for allergen content by immunoaffinity capillary elecrophoresis-matrix assisted laser desorption/ionization mass spectrometry, as well as a simplified version of this technique, the immunomagnetic separation -matrix-assisted laser desorption/ionization mass spectrometry.

Visit 2 (V2): During this visit, the parents/patients will report on the brand, the frequency and the amount of "may contain" foods eaten since V1.

The quality of life questionnaire will be filled out again by the parents/patient.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-18 years at time of inclusion
* Tree nut or peanut allergy documented by:

  * Positive skin prick tests (SPTs) to peanut and/or tree nuts
  * Positive specific IgE (sIgE) to peanut and/or tree nuts ( ≥0.35 kU/L)
  * A recent (< 1 year) positive food challenge, reacting to the dose of 30 mg of proteins or below.
* Parent/Legal guardian has been informed about the study and has signed Informed Consent Form

Exclusion Criteria:

* History of a moderate or severe reaction during a food challenge with a dose of 30 mg of proteins or less.
* Expected non-adherence to the study protocol.
* Severe or uncontrolled asthma.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Result of the food challenges with foods labelled with "may contain traces" (tolerated or reacted). | At study entry
  Result of the food challenges with foods labelled with "may contain traces" (tolerated or reacted).

SECONDARY OUTCOMES:
Tolerance to foods labelled with "may contain traces" eaten normally during a 3 months follow-up. | During 3 months follow-up
  Tolerance to foods labelled with "may contain traces" eaten normally during a 3 months follow-up (reactions / no reactions to these foods).
Frequency of reactions to foods labelled with "may contain traces" eaten normally during a 3 months follow-up. | During 3 months follow-up
  Frequency of reactions to foods labelled with "may contain traces" eaten normally during a 3 months follow-up (number of reactions).
Severity of reactions to foods labelled with "may contain traces" eaten normally during a 3 months follow-up. | During 3 months follow-up
  Severity of reactions to foods labelled with "may contain traces" eaten normally during a 3 months follow-up (severity of reactions by reaction type).
Changes of quality of life after 3 months without restriction of foods labelled with "may contain traces", compared to baseline when restricting. | At entry and after 3 months
  Changes of quality of life measured with the age-appropriate "Food allergy quality of life questionnaire (0-12 years [parents], 7-12 years [patients], or 13-17 years [patients]. Results (on a continuous numerical ranking from 1 to 6 for each item) after 3 months without restriction of foods labelled with "may contain traces", are compared to baseline when restricting.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Eigenmann, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Pediatric Allergy Unit - University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No